CLINICAL TRIAL: NCT05119894
Title: A Multicenter, Open-label, Clinical Pharmacology Trial to Determine the Pharmacokinetics, Tolerability, and Safety of Brexpiprazole Long Acting Injectable (LAI) Administered as a Single Dose in Patients With Schizophrenia
Brief Title: A Clinical Pharmacology Trial of Brexpiprazole Long Acting Injectable (LAI) Administered as a Single Dose in Patients With Schizophrenia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision:Change the Development plan
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 331-102-00373; jRCT2061210051 (Other: jRCT)
Record Dates: First submitted 2021-11-12; First posted 2021-11-15 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Brexpiprazole LAI: Dose 1 (Experimental)
  Interventions: Drug: Brexpiprazole LAI: Dose 1
- Brexpiprazole LAI: Dose 2 (Experimental)
  Interventions: Drug: Brexpiprazole LAI: Dose 2
- Brexpiprazole LAI: Dose 3 (Experimental)
  Interventions: Drug: Brexpiprazole LAI: Dose 3
- Brexpiprazole LAI: Dose 4 (Experimental)
  Interventions: Drug: Brexpiprazole LAI: Dose 4

INTERVENTIONS:
Drug: Brexpiprazole LAI: Dose 1 — Cohort 1: Single Dose Intramuscular Injection: Brexpiprazole LAI Dose 1
  Arms: Brexpiprazole LAI: Dose 1
Drug: Brexpiprazole LAI: Dose 2 — Cohort 2: Single Dose Intramuscular Injection:Brexpiprazole LAI Dose 2
  Arms: Brexpiprazole LAI: Dose 2
Drug: Brexpiprazole LAI: Dose 3 — Cohort 3: Single Dose Intramuscular Injection:Brexpiprazole LAI Dose 3
  Arms: Brexpiprazole LAI: Dose 3
Drug: Brexpiprazole LAI: Dose 4 — Cohort 4: Single Dose Intramuscular Injection:Brexpiprazole LAI Dose 4
  Arms: Brexpiprazole LAI: Dose 4

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (PK), tolerability and safety of brexpiprazole LAI following a single administration in subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients who are between 18 and 64 years of age, inclusive, at the time of informed consent
* Patients with a diagnosis of schizophrenia as defined by the DSM-5® criteria
* Patients who are able to remain at the trial site for the protocol-defined hospitalization period
* Patients with a body mass index [BMI = body weight (kg) / height (m)2] of no less than 18.5 kg/m2 and less than 35.0 kg/m2 at screening
* Patients who are able to provide written informed consent (if the patient is a minor or is hospitalized for medical protection, his or her legally acceptable representative must also give informed consent) prior to commencement of any trial procedure and are judged by the investigator or subinvestigator to be able to meet all protocol-defined requirements

Exclusion Criteria:

* Patients with a diagnosis of a concurrent mental disorder besides schizophrenia (eg, schizoaffective disorder, major depressive disorder, bipolar I disorder, bipolar II disorder, general anxiety disorder, obsessive-compulsive disorder, post-traumatic stress disorder, dementia or mild neurocognitive disorder, and personality disorder) as defined by the DSM-5® criteria. However, this exclusion does not apply to caffeine- or tobacco-related disorders.
* Patients who fail to meet the mandatory washout periods for the prohibited concomitant drugs and foods before commencement of IMP administration, or patients who are anticipated to take any of the drugs or foods during the trial period
* Patients who have received electroconvulsive therapy (ECT) within 60 days prior to the administration of IMP
* Patients with clinically significant nervous, hepatic, renal, metabolic, blood, immune, cardiovascular, respiratory, or digestive system disorders However, such patients may be enrolled if the condition is mild or well controlled and is considered to not affect safety or PK evaluations.
* Patients who have met the DSM-5® diagnostic criteria for substance-related or addictive disorder, including alcohol and benzodiazepines but excluding caffeine and tobacco, within 180 days prior to the administration of IMP
* Patients with a positive drug test at screening (according to the results from the central laboratory). However, such patients may be enrolled if their condition is not diagnosed as a substance-related or addictive disorder, according to the DSM-5® diagnostic criteria.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of brexpiprazole | Blood Sampling for plasma drug measurement Day 1 (predose and 4, 8, 12 hours postdose), 2, 3, 5,7,9,11,13,15,17,19, 21, 25, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91, 98, 112, 126, 154, 182

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.